CLINICAL TRIAL: NCT06896513
Title: Relationship of Isthmus Thickness With Difficult Laryngoscopy and Difficult Intubation in Patients Receiving Hypothyroidism Treatment: A Prospective Observational Clinical Study
Brief Title: Relationship of Isthmus Thickness With Difficult Laryngoscopy and Difficult Intubation in Patients Receiving Hypothyroidism Treatment
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Ömer Keklicek, Principal Investigator MD, Konya City Hospital
Other Study IDs: 2024/5150
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-04

CONDITIONS: Difficult Intubation; Difficult Laryngoscopy
Keywords: Intubation; Laryngoscopy; Isthmus
MeSH Terms: interventions — pax2a protein, zebrafish

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients with known hypothyroidism who are receiving medical treatment and are scheduled for e: Adult patients with known hypothyroidism who are receiving medical treatment and are scheduled for elective intubation.
  Interventions: Other: Isthmus

INTERVENTIONS:
Other: Isthmus — The neck skin thickness from the thyroid isthmus to the skin will be measured in millimeters using a linear ultrasound probe (3-13 Hz) in the supine position with neck hyperextension. Measurements will be taken in a transverse view at the level of the 2nd-3rd tracheal rings, and the average of three measurements will be recorded.

SUMMARY:
Under general anesthesia, the rate of failed intubation ranges from 1.5% to 13%, raising concerns among anesthesiologists whose primary goal is successful airway management. In this context, various physical and ultrasonographic measurement techniques have been developed to predict difficult intubation. Ultrasonography is effectively used for estimating tracheal tube size, device placement, diagnosing upper airway pathologies, and guiding percutaneous tracheostomy. In thyroid pathologies, intubation difficulty may increase; however, the impact of goiter remains debatable, as some conditions causing hypothyroidism are reported to lead to thyroid gland atrophy rather than hypertrophy. The study's hypothesis is that an atrophic or fibrotic thyroid isthmus may be associated with difficult laryngoscopy and intubation. Evaluation will be performed using the Cormack-Lehane score (Grade III-IV) and the Intubation Difficulty Scale (IDS >5). The aim is to determine the relationship between thyroid isthmus thickness and difficult laryngoscopy and intubation during elective intubation in patients receiving hypothyroidism treatment.

Preoperatively, patients' demographic and clinical data (age, gender, height, weight, BMI, comorbidities, ASA score, thyroid medication dose, treatment duration, and type of thyroid disease) will be recorded. In the premedication room, after administering 0.01 mg/kg IV midazolam, the distance between the thyroid isthmus and the skin will be measured using a linear ultrasound probe (3-13 Hz) in the supine position with neck hyperextension at the level of the 2nd-3rd tracheal rings; the average of three measurements will be recorded. In the operating room, under noninvasive monitoring and following mask pre-oxygenation, anesthesia induction will be performed using IV 2 mg/kg propofol, 1 µg/kg fentanyl, 1 mg/kg lidocaine, and 0.6 mg/kg rocuronium. Once the TOF reaches zero, an experienced anesthesiologist will intubate using a size 3 Macintosh blade for females and size 4 for males with an appropriate endotracheal tube. The intubation time, defined as the interval from laryngoscope insertion until the first capnography wave is detected, will be recorded along with the Cormack-Lehane and EZS scores and the requirement for video laryngoscopy. In cases of failed intubation, the 2022 ASA Difficult Airway Management Guidelines will be applied.

DETAILED DESCRIPTION:
Under general anesthesia, the rate of failed intubation ranges between 1.5% and 13%, a high rate that raises concerns among anesthesiologists whose primary objective is successful airway management. Consequently, various physical examination and ultrasonographic measurement methods have been developed to predict difficult intubation. While anesthesiologists previously relied on bedside physical examinations, the widespread availability, reliability, and portability of ultrasound (USG) have promoted its use in airway evaluation. USG is used to assess the difficult airway, estimate tracheal tube size, ensure proper placement of the tracheal tube and laryngeal mask, diagnose upper airway pathologies, and guide percutaneous tracheostomy.

In thyroid pathologies, intubation difficulty may increase. Although difficult intubation rates in thyroid surgery-a known risk factor-range from 6.8% to 9.6%, some studies suggest that the presence of a goiter is not associated with difficult intubation. The literature has mostly examined the relationship between intubation difficulty and hypertrophic thyroid tissue; however, certain conditions causing hypothyroidism (e.g., Hashimoto's thyroiditis and atrophic thyroiditis) may lead to thyroid gland atrophy. Our hypothesis is that an atrophic or fibrotic thyroid isthmus is (or is not) associated with difficult laryngoscopy and intubation.

Difficult laryngoscopy is defined as the inability to visualize the vocal cords despite multiple laryngoscopic attempts. Tracheal intubation that requires multiple attempts or fails after several attempts is termed difficult or failed intubation. Evaluation will be performed using the Cormack-Lehane (C&L) score and the Intubation Difficulty Scale (IDS). The C&L score classifies the laryngeal view into four grades based on the visualization of the vocal cords and epiglottis (Grade I: full view of the glottis; Grade II: partial view; Grade III: only the epiglottis is visible; Grade IV: neither the epiglottis nor the glottis is visible), with Grades III-IV being associated with difficult laryngoscopy. The IDS, which consists of seven parameters, indicates a difficult airway when the score exceeds 5. Accordingly, a C&L classification of Grade III-IV and an IDS >5 will be considered indicative of difficult laryngoscopy and intubation.

The primary aim of this study is to determine the relationship between thyroid isthmus thickness and difficult laryngoscopy and intubation during elective intubation in patients receiving hypothyroidism treatment. The primary hypothesis is that an atrophic or fibrotic thyroid isthmus is associated with difficult laryngoscopy and intubation, while the secondary hypothesis posits that the duration of hypothyroidism treatment is associated with difficult laryngoscopy and intubation.

This study will include adult patients with known hypothyroidism who are undergoing surgery for any reason at Konya City Hospital and are receiving medical treatment, with an ASA score of 2-3. Patients will be excluded if they have a known history of difficult intubation, a body mass index (BMI) >40, airway pathology, conditions that restrict neck movements (e.g., rheumatoid arthritis, systemic lupus erythematosus, ankylosing spondylitis), a cervical range of motion ≤80°, a history of cervical radiotherapy, or if they do not consent to participate. The primary objective is to evaluate the efficacy of thyroid isthmus muscle thickness in predicting difficult intubation in goiter patients undergoing thyroidectomy.

Preoperatively, patients' age, gender, height (cm), weight (kg), BMI, comorbidities, ASA score, thyroid medication dose, duration of hypothyroidism treatment (years), and type of thyroid disease (Hashimoto's thyroiditis, atrophic thyroiditis, multinodular goiter, malignant goiter) will be recorded. In the premedication room, after administering 0.01 mg/kg IV midazolam, the neck skin thickness from the thyroid isthmus to the skin will be measured in millimeters using a linear ultrasound probe (3-13 Hz) in the supine position with neck hyperextension. Measurements will be taken in a transverse view at the level of the 2nd-3rd tracheal rings, and the average of three measurements will be recorded.

In the operating room, patients will be monitored using noninvasive blood pressure, pulse oximetry, electrocardiography, bispectral index (BIS), and neuromuscular monitoring (TOF). Following mask pre-oxygenation, anesthesia induction will be performed with IV 2 mg/kg propofol, 1 µg/kg fentanyl, 1 mg/kg lidocaine, and 0.6 mg/kg rocuronium. Once the TOF value reaches zero, an experienced anesthesiologist will intubate the patient using an appropriately sized endotracheal tube with a size 3 Macintosh blade for females and a size 4 for males, following proper head positioning. The intubation time-defined as the interval from laryngoscope insertion until the first capnography waveform is detected-will be recorded. Additionally, the patients' Cormack-Lehane and IDS scores, as well as the need for video laryngoscopy, will be documented. In the event of failed intubation, management will be conducted in accordance with the 2022 ASA Difficult Airway Management Guidelines (e.g., summoning assistance, optimizing oxygenation, selecting an invasive or noninvasive approach, considering combination techniques, limiting the number of intubation or supraglottic airway placement attempts to prevent potential injury and complications, ensuring that any invasive airway procedure is performed by a trained individual as rapidly as possible, and initiating ECMO when appropriate/available).

ELIGIBILITY:
Inclusion Criteria:

* Known hypothyroidism receiving medical treatment
* ASA score of 2-3

Exclusion Criteria:

* Known history of difficult intubation
* Body mass index (BMI) > 40
* Presence of airway pathology
* Diseases that restrict neck movement (e.g., RA, SLE, AS, etc.)
* Head and neck range of motion ≤ 80°
* History of cervical radiotherapy
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery at Konya City Hospital for any reason Known hypothyroidism receiving medical treatment
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Cormack-Lehane score and Intubation Difficulty Scale values of patients whose isthmus thickness is below 3 mm. | From enrollment to the end of treatment at 6 Mounths

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol